CLINICAL TRIAL: NCT01346098
Title: Total Pancreatectomy With Islet Autotransplantation as a Superior Alternative to Pancreatoduodenectomy in Patients at Very High-risk of Complications of the Pancreatic Anastomosis: a Single-center Prospective Randomised Clinical Trial
Brief Title: Islet Autotransplantation in Patients at Very High-risk Pancreatic Anastomosis
Acronym: PAN-IT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Ministry of education, university and research, Italy (Unknown)
Responsible Party: Principal Investigator, Piemonti Lorenzo, Director Islet Transplantation Program, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAN-IT
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Postpancreatectomy Hyperglycemia
Keywords: diabetes; islet transplantation; pancreas; pancreatectomy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP B (Experimental): At the time of surgery the surgeon will directly assess pancreatic consistency and the pancreatic duct size. In the presence of a soft pancreas and a small duct (diameter <3 mm), the patient will be randomly assigned to receive either a pancreaticoduodenectomy with pancreatic anastomosis (group A) or a total pancreatectomy with IAT (group B).
  Interventions: Procedure: Total pancreatectomy with islet autotransplantation
- GROUP A (Active Comparator)
  Interventions: Procedure: Pancreaticoduodenectomy with pancreatic anastomosis

INTERVENTIONS:
Procedure: Pancreaticoduodenectomy with pancreatic anastomosis — Standard lymphadenectomy, end-to-side two-layer pancreaticojejunostomy and duodenojejunostomy will be performed. If the pylorus is preserved, so will be the right gastric artery, unless the artery is damaged or hindering adequate gastric mobilization. No prokinetic agent will be administered routinely, but IV metoclopramide will given on demand (10 mg , three times daily). Prophylaxis will consist of octreotide (0,1 mg three times daily from day 0 to 7), low molecular weight heparin and a single dose of antibiotic (cefazolin 2 g). Early postoperative analgesia will be achieved by epidural or, when contraindicated, patient-controlled analgesia
  Arms: GROUP A
Procedure: Total pancreatectomy with islet autotransplantation — If the patient will be assigned to this group, the surgeon will complete the pancreatectomy preserving the spleen. The body and tail of the pancreas will be sent to the islet isolation facility. Islets will be isolated and purified according to the automated method described by Ricordi. The resulting islet tissue will be suspended in a cold isotonic saline solution and infused into the portal vein during the next 24h.
  Arms: GROUP B

SUMMARY:
The goal of the proposal is to demonstrate that, in patients with disease of the pancreatic head with very high-risk of complications of pancreatojejunal reconstruction (soft pancreas and pancreatic duct diameter <3 mm), total pancreatectomy with islet autotransplantation (IAT) is associated with a lower morbidity (in terms of surgical or medical complications) and mortality compared with pancreaticoduodenectomy and pancreatojejunal anastomosis.

DETAILED DESCRIPTION:
Complications of the pancreatic anastomosis still represents a significant risk for death after the resection of the pancreatic head. In an effort to decrease morbidity and mortality, the referral of patients who need a pancreaticoduodenectomy to institutions (and surgeons) performing a high volume of this surgical procedure has been championed. Nonetheless, the role of prophylactic medications and the best surgical technique(s) for the removal of the pancreatic head are still debated. However, very few prospective randomized clinical trials have been conducted to compare different surgical techniques.

Our study will address for the first time the role for preemptive total pancreatectomy and IAT in selected patients undergoing pancreaticoduodenectomy that are considered high risk for pancreaticojejunostomy disruption (eg, small pancreatic duct, soft pancreas). The information expected is the identification of total pancreatectomy and the IAT as the standard treatment in a subgroup of patient with pathologies of the pancreatic head at high risk for leakage of pancreatic anastomosis. Ultimately this project will lead to reserve more innovative cell therapy for patients with the highest risk of anastomosis failure reducing pancreatojejunal reconstruction related morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Ability to provide written informed consent
* Mentally stable and able to comply with the procedures of the study protocol
* Fasting glycaemia <126 mg/dl without glucose-lowering medications.

Exclusion Criteria:

* Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial
* Diagnosis of intraductal papillary mucinous cancer, unless the absence of multifocal lesion is demonstrated by endoscopic US
* Presence of multifocal or residual disease at the pancreatic margin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
incidence of complications after pancreatic surgery | 90 days from discharge
  Complications will be defined and graded according to the Novel Grading System classification ( DeOliveira et al 2006). A special emphasis is given to life-threatening and permanently disabling complications.

SECONDARY OUTCOMES:
Incidence of each individual postoperative complication | 90 days from discharge
  1. death
  2. pancreatic fistula defined according to the International Study Group on Pancreatic Fistula (Bassi C et al 2005)
  3. delayed gastric emptying (DGE) defined according to the International Study Group on Pancreatic Fistula (Wente et al 2007)
  4. intra-abdominal complications
  5. medical complications
Incidence of endocrine and exocrine pancreatic insufficiency | 12 months after surgery.
  We will assess endocrine pancreatic function by measuring fasting plasma glucose and HbA1c in all patients.
  Clinical hallmarks of pancreatic exocrine insufficiency include symptoms of fat malabsorption, such as steatorrhea, weight loss and abdominal pain. Frequency of bowel movements and characteristics of stools will be serially recorded. Fat-soluble vitamins such as A, D, E and K will be measured 12 month after the hospital discharge after the index surgery. Oral pancreatic enzyme supplementation will be prescribed according to the severity of clinical steatorrhea and weight loss.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Fondazione Centro San Raffaele del Monte Tabor; Gianpaolo Balzano, MD, Study Director — Fondazione Centro San Raffaele del Monte Tabor
Locations (1):
- IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Balzano G, Zerbi A, Aleotti F, Capretti G, Melzi R, Pecorelli N, Mercalli A, Nano R, Magistretti P, Gavazzi F, De Cobelli F, Poretti D, Scavini M, Molinari C, Partelli S, Crippa S, Maffi P, Falconi M, Piemonti L. Total Pancreatectomy With Islet Autotransplantation as an Alternative to High-risk Pancreatojejunostomy After Pancreaticoduodenectomy: A Prospective Randomized Trial. Ann Surg. 2023 Jun 1;277(6):894-903. doi: 10.1097/SLA.0000000000005713. Epub 2022 Sep 30. PMID 36177837